CLINICAL TRIAL: NCT00309413
Title: A Placebo-Controlled Randomized Cross-Over Clinical Trial on the Antipsychotic Properties of the Endocannabinoid Modulator Cannabidiol
Brief Title: A Clinical Trial on the Antipsychotic Properties of Cannabidiol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Stanley Medical Research Institute (Other); Coordinating Centre for Clinical Trials Cologne (Other)
Responsible Party: F. Markus Leweke, M.D., University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-PT 04-153
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia and Disorders with Psychotic Features
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cannabidiol/Placebo
  Interventions: Drug: Cannabidiol/Placebo
- 2 (Placebo Comparator): Placebo/Cannabidiol
  Interventions: Drug: Placebo/Cannabidiol

INTERVENTIONS:
Drug: Placebo/Cannabidiol — 600 mg/day, oral, capsules, 2 weeks, than cross-over
  Arms: 2
Drug: Cannabidiol/Placebo — 600 mg/day, oral, capsules, 2 weeks, than cross-over
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether cannabidiol, a herbal cannabinoid, is effective in the treatment of acute schizophrenic or schizophreniform psychosis in a placebo-controlled, randomized double-blind study.

DETAILED DESCRIPTION:
Despite recent advances in the treatment of schizophrenia and schizophreniform disorders, there is still a need to develop efficient and better tolerated psychopharmacological approaches to this group of diseases. The endogenous cannabinoid system provides a promising target in the pharmacotherapy of these disorders. This approach is based upon recent findings indicating that the human endogenous cannabinoid system is significantly involved in the pathogenesis of schizophrenia and that cannabidiol is effective in treating acute psychotic symptoms of schizophrenic patients. We will investigate cannabidiol versus placebo in a randomized, double blind design with extensive safety measures.

The primary hypothesis to be tested is that Cannabidiol is expected to be superior to placebo in the treatment of acute schizophrenic and schizophreniform psychoses with regard to its antipsychotic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Diagnosis of schizophrenic or schizophreniform psychosis
* Minimal initial score of 36 in the BPRS total score and a minimum of 12 in the BPRS Psychosis Cluster, including items 4 (conceptional disorganisation), 8 (exaggerated self-esteem), 12 (hallucinatory behaviour), and 15 (unusual thought content)
* Exclusion of pregnancy in female subjects through negative β-HCG test

Exclusion Criteria:

* Lack of accountability
* Pregnancy or risk of pregnancy or lactation.
* Other relevant interferences of axis 1 according to diagnostic evaluation through MINI including undifferentiated residual forms of schizophrenia.
* Treatment with depot-antipsychotics during the last three months.
* Severe internal or neurological illness, especially cardiovascular, renal, advanced respiratory, haematological or endocrinological failures. Positive Hepatitis-serology.
* QTc-elongation.
* Acute suicidal tendency of or hazard to others by the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
BPRS | 2 x 2 weeks

SECONDARY OUTCOMES:
PANSS, EPS, Prolactin, ECG etc. | 2 x 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Dept. of Psychiatry and Psychotherapy, Cologne, North Rhine-Westphalia, Germany